CLINICAL TRIAL: NCT06119399
Title: Effect Of Diaphragmatic Doming Versus Breathing Exercises On Ventilatory Function And Core Endurance In Chronic Neck Pain Patients
Brief Title: Diaphragmatic Doming vs Breathing Exercises on Ventilatory Function & Core Endurance in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mina Atef Georgui Elias (Other)
Responsible Party: Sponsor-Investigator, Mina Atef Georgui Elias, Lecturer of Internal Medicine and Geriatric, Faculty of Physical Therapy, Badr University in Cairo., Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003656
Record Dates: First submitted 2023-10-28; First posted 2023-11-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
Keywords: Chronic Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises Plus Conventional Exercise Program for Chronic Neck Pain (Experimental): Subjects will receive conventional exercise program for Chronic Neck Pain in addition to breathing exercises (diaphragmatic and pursed lip breathing) for (three sessions per week for six weeks).
  Interventions: Other: Diaphragmatic Breathing Exercise; Other: Pursed Lip Breathing Exercise; Other: Conventional exercise program for chronic neck pain
- Doming of the diaphragm plus Conventional Exercise Program for Chronic Neck Pain (Experimental): Patients in this arm will receive conventional physiotherapy treatment for Chronic Neck Pain in addition to doming of the diaphragm (three sessions per week for six weeks).
  Interventions: Other: Doming of the diaphragm; Other: Conventional exercise program for chronic neck pain

INTERVENTIONS:
Other: Diaphragmatic Breathing Exercise — Diaphragmatic breathing exercise will be taught by placing the subject comfortably positioned with either therapist or the patient's hand directed over the abdominal area and instructing the subjects to focus on an outward movement of the abdominal area throughout inspiration and an inward movement of the abdominal area during expiration. (4 sets, and as each set had 4 complete breathing breaks, these exercises will be conducted for 3 days a week for 6 weeks)
  Arms: Breathing Exercises Plus Conventional Exercise Program for Chronic Neck Pain
Other: Pursed Lip Breathing Exercise — Pursed lip breathing exercises will be performed by necessitating the subjects to inhale through their nose and then exhaling slowly for a period of 4-6 s by pursing the lips
  Arms: Breathing Exercises Plus Conventional Exercise Program for Chronic Neck Pain
Other: Doming of the diaphragm — * The physiotherapist places the thumbs just inferior to the patient's lower costal margin and xiphoid process with the thumbs pointing cephalad.
  * The patient is instructed to take a deep breath and exhale. On exhalation, the physiotherapist's thumbs follow the diaphragm, which permits the thumbs to move posteriorly.
  * The patient is instructed to inhale, and the physiotherapist gently resists this motion.
  * The patient is instructed to exhale, and the physiotherapist gently follows this motion posteriorly and cephalad, as the thumbs are now beneath the costal margin and xiphoid process.
  * The patient inhales as the physiotherapist maintains pressure on the upper abdomen and then, on repeated exhalation, encourages further cephalad excursion.
  * This procedure is repeated for three to five respiratory cycles until the diaphragm domes easily at the end of exhalation.
  Arms: Doming of the diaphragm plus Conventional Exercise Program for Chronic Neck Pain
Other: Conventional exercise program for chronic neck pain — Patients will perform three repetitions of stretching exercises for neck flexor, extensor, lateral flexor, and rotator for 30 seconds as warm-up and cool-down exercises, to relieve tension on each side of the neck.
  Then cranio-cervical flexion exercise will be started using feedback from an air-filled pressure sensor placed behind the neck. Subjects will lay in the crook lying position. The pressure biofeedback unit will be placed below the occiput and inflated up to a baseline pressure of 20 mmHg. The subjects will be instructed to perform head-nodding action to progressively target 5 pressure levels (hold 10 seconds with brief rest periods between each contraction 3-5 seconds). This includes 3 sets in a session for 10 repetitions each with 2 minutes of rest between sets and 3days a week for 6 weeks.

SUMMARY:
The purpose of the study is to investigate if there is any difference between effect of diaphragmatic doming versus breathing exercises on ventilatory function and core endurance in patients with chronic neck pain

DETAILED DESCRIPTION:
Patients with chronic neck pain will be participated in this comparative study.

They will be divided into 2 groups:

Group (A) will be consisted of 30 patients who will receive conventional physiotherapy treatment for chronic neck pain plus breathing exercise (diaphragmatic and pursed lip breathing) (Three sessions per week for 6 weeks) Group (B) will be consisted of 30 patients who will receive conventional physiotherapy treatment for chronic neck pain plus Doming of the diaphragm (Three sessions per week for 6 weeks)

Pulmonary functions and neck endurance will be assessed for all patients in both groups before the first session and after the last session

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic neck pain (for more than 3 months)
* Their age ranged from 20 to 30 years old
* Their body mass index ranged from (18.5 -29.9) kg/m2
* Poor results on the cranio-cervical flexion (CCF) test using a pressure biofeedback instrument.

Exclusion Criteria:

* History of respiratory disease and Clinical signs of a severe cardiac event.
* Severe psychiatric or cognitive impairment
* Tumor and Spinal fractures
* Spinal cord compression that required urgent surgery
* Current or past Smokers
* Obese (BMI >30) or underweight (BMI ˂18.5)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Endurance of deep cervical flexors | 6 weeks
  Endurance of deep cervical flexors muscles will be measured by the cranio-cervical flexion test using a pressure biofeedback instrument.
  During the cranio-cervical flexion test, the subject lay in the crook lying position and the pressure biofeedback instrument will be placed under the neutral cervical spine below the occiput and inflated up to 20 mmHg.
  The subjects will perform this movement at 5 different pressure levels, i.e., 22, 24, 26, 28, and 30 mmHg. Each level will be supposed to be held for 10 s, and the test will be terminated if they were unable to hold the position for 10 s at any level or if the maximum level was achieved (30 mmHg).
Forced expiratory volume in the first second (FEV1) | 6 weeks
  Forced expiratory volume in the first second (FEV1) is one of ventilatory function test parameters, measured using Spirometry, Model SpirOx plus (by Meditech company-China)
  The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
Forced vital capacity (FVC). | 6 weeks
  Forced vital capacity (FVC) is one of pulmonary function test parameters, measured using Spirometry, Model SpirOx plus (by Meditech company-China)
  Forced vital capacity (FVC) is the volume of air that can forcefully expired from the lungs following maximum inspiration, it is measured in liters.
Peak expiratory flow rate (PEFR) | 6 weeks
  Peak expiratory flow rate (PEFR) is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration, measured in liters per second.
  Peak expiratory flow rate (PEFR) as a pulmonary function, is measured using Spirometry, Model SpirOx plus (by Meditech company-China)
Neck Disability Index (NDI) | 6 weeks
  Neck function is assessed using the self-reported Neck Disability Index (NDI), which is a valid and reliable test for measuring neck disability. The NDI consists of 10 items referring to daily activities (work, lifting, driving, sleeping, reading, headaches, recreation, concentration, personal care, and pain intensity). Each item (ranging from 0 to 5, with a score of 0 for no pain and no limitation and a score of 5 for maximum pain and limitation). The total maximum score is 50.
Visual Analogue Score for pain intensity | 6 weeks
  Visual Analogue score is a measure of pain severity, it is assessed by the self-reported Visual Analogue Scale (VAS).
  The Visual Analogue Scale evaluates the intensity of pain. It consists of a 10 cm line, that has two end points, where 0 represents "no pain at all" while 10 indicates "most severe pain".
  Every patient is asked to rate his/her level of pain by placing a mark on the line. Use a ruler to measure the distance in centimetres from the 'no pain' (or zero) to the current pain mark.
  This provides pain intensity score out of 10.

SECONDARY OUTCOMES:
FEV1/FVC ratio | 6 weeks
  FEV1/FVC ratio is a calculated ratio of Forced expiratory volume in the first second (FEV1) to Forced vital capacity (FVC).
  t represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).

CONTACTS AND LOCATIONS:
Overall Officials: Eman NE Sayed, M.Sc., Principal Investigator — Assistant Lecturer, dept of internal medicine & geriatric, Badr University in Cairo.; Mina AG Elias, Dr., Study Chair — Lecturer, dept of internal medicine & geriatric, Badr University in Cairo.; Hany E Obaya, Ass.Prof.Dr, Study Director — Dept of PT for Cardiovascular/Respiratory Disorder & Geriatrics, Faculty of PT, Cairo Univ.; Asmaa M Sharabash, Dr., Study Chair — Dept of PT for Cardiovascular/Respiratory Disorder & Geriatric, Faculty of PT, Cairo Univ.
Locations (2):
- Egypt (2):
  - Outpatient Clinic; Faculty of Physical Therapy, Badr University in Cairo., Cairo, Badr
  - Outpatient clinic, Faculty of physical therapy, Cairo University., Giza, Dokki

IPD SHARING:
Plan to Share IPD: No